CLINICAL TRIAL: NCT06001242
Title: Voleybolcularda Üst Ekstremite Patlayıcı Güç Ile Gövde Kaslarının Arasındaki İlişkinin İncelenmesi
Brief Title: The Relationship Between Upper Extremity Explosive Power and Trunk Muscles in Volleyball Players
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: GO 23/540
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Ultrasonography; Upper Extremity; Physical Endurance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Volleyball is an interval sport involving consecutive aerobic and anaerobic loads. Strength training based on explosive movements can improve performance in the upper extremities. Strength performance has an important place in this sport. Trunk stabilization is defined as 'proximal stability for distal mobility'. Disorder in any segment of the kinetic chain model will affect the quality of movement in the lower and upper segments.The aim of this study is to examine the relationship between the morphological features of the transversus abdominis, lumbal multifidus (L4-5), internal external oblique muscles, and the anaerobic power of the upper extremity and shoulder girdle functionThis study was designed as a cross-sectional. They will consist of 30 volleyball players between 14-30 years of age. Muscle morphological features of the participants by ultrasound; explosive strength will be evaluated by Medicine Ball Throw test, functional evaluation will be evaluated by Closed Kinetic Chain Upper Extremity Endurance test.

ELIGIBILITY:
Inclusion Criteria:

* Training for an hour at least 3 days a week for at least 1 year
* Body Mass Index (BMI) below 30 kg/m2
* No concomitant neurological, rheumatological or systemic disease
* Volunteer to participate in the study.

Exclusion Criteria:

* Having any surgery / serious pathology of the spinal column
* Having had an upper extremity injury in the last 6 months that would affect his ability to play volleyball
* Having an injury that requires at least 2 weeks of discontinuation
* Severe musculoskeletal/systemic discomfort during the measurements.

Ages: 14 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Hacettepe University will be directed from the referred athletes
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-26 (Estimated); Primary Completion 2025-08-26 (Estimated); Study Completion 2025-08-26 (Estimated)

PRIMARY OUTCOMES:
Muscle morphology | 1 day
  Morphological characteristics transverse abdominis, lumbar multifidus,internal obliquus, external obliquus will be evaluated via ultrasound imaging

SECONDARY OUTCOMES:
Expolsive Power | 1 day
  Medicine Ball Throw
Core stability | 1 day
  Sharmannn's Core Stability Test
Upper Extremity Endurance | 1 day
  Closed Kinetic Chain Upper Extremity Stability Test

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Aynur Demirel, Ankara, Turkey (Türkiye)